CLINICAL TRIAL: NCT05557903
Title: Recombinant Humanized Anti-CD52 Monoclonal Antibody in the Treatment of Relapsed and Refractory NHL and Initially Treated T-PLL Phase I Clinical Study on Safety and Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy
Brief Title: Phase Ⅰ Clinical Study of Anti-CD52 Monoclonal Antibody in NHL and T-PLL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RD04-CD52-V01
Record Dates: First submitted 2022-02-19; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, T-Cell
Keywords: anti-CD52 monoclonal antibody; relapsed and refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Recurrence | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group of anti-CD52 monoclonal antibody (Experimental): safety and tolerability, pharmacokinetic characteristics and preliminary efficacy in the treatment of relapsed and refractory nhl (including cll/sll, pll, ptcl, diffuse large b-cell lymphoma, follicular cell lymphoma, mantle cell lymphoma, and marginal zone lymphoma) and initially treated t-pll of recombinant humanized anti-cd52 monoclonal antibody injection
  Interventions: Biological: Recombinant Humanized Anti-CD52 Monoclonal Antibody Injection

INTERVENTIONS:
Biological: Recombinant Humanized Anti-CD52 Monoclonal Antibody Injection — Single dosing: DLT observation for 7 days after administration; Multiple dosing: 3times/weeks,12 times, 28 days of DLT observation
  Other Names: Anti-CD52 Monoclonal Antibody

SUMMARY:
Phase I clinical study of multicenter, single-arm, open, non-randomized evaluation of recombinant humanized anti-CD52 monoclonal antibody in the NHL and T-PLL

DETAILED DESCRIPTION:
Recombinant Humanized Anti-CD52 Monoclonal Antibody Injection in the Treatment of Relapsed and Refractory NHL (Including CLL/SLL, PLL, PTCL, Diffuse Large B-cell Lymphoma, Follicular Cell Lymphoma, Mantle Cell Lymphoma, and Marginal Zone Lymphoma) and Initially Treated T-PLL Phase I Clinical Study on Safety and Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy

ELIGIBILITY:
Inclusion Criteria:

For Patients With Relapsed And Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma/Lymphoblastic Leukemia (CLL/SLL/PLL) And Initial Treated t-Lymphoblastic Leukemia ( InitialTreated T-PLL)

-Patients with CLL/SLL or PLL were confirmed by histopathological or flow immunotyping;

1. Patients with indications for treatment according to iwCLL2018 criteria and determined by the investigator;
2. Age from 18 to 70 (including boundary value), no gender limitation;
3. ECOG physical condition score 0 ~ 2;
4. Patients have measurable lesions (lymphadenopathy (maximum baseline diameter ≥1.5 cm), or hepatomegaly/splenomegaly due to CLL or PLL or peripheral tumor lymphocytes >5×10E9/L);
5. CLL/SLL patients are intolerant or resistant to previous BTK inhibitor treatment; Or newly treated patients with T-PLL; Or relapse-resistant PLL (relapse-resistant PLL is defined as disease progression following recent remission of treatment. Treatment-resistant disease was defined as failure to achieve ≥PR from the most recent treatment or disease progression within 6 months of the last treatment);
6. Laboratory test results must meet the following requirements (no blood components, short-acting cell growth factor and other drugs are allowed within 7 days prior to laboratory test; Long-acting growth factor is not allowed within the first 14 days), and laboratory test results within 7 days before screening;

   * Bone marrow function: Neutrophils ≥1×10E9/L, platelets ≥50×10E9/L, and hemoglobin ≥75g/L were observed without growth factor support treatment.
   * Liver function: AST and ALT ≤2×ULN (no liver invasion); Alanine aminotransferase or/and aspartate aminotransferase ≤5×ULN (liver aggressor). Total bilirubin ≤2×ULN;
   * Renal function: serum creatinine ≤2×ULN and creatinine clearance rate > 50mL/min;
   * Blood coagulation function: international standardized ratio (INR) ≤1.5×ULN and activated partial thrombin time (APTT) ≤1.5×ULN;
7. Life expectancy > 3 months;
8. Fertile men and women of reproductive age are willing to take effective contraceptive measures from the signing of informed consent to 6 months after the last administration of the experimental drug; Women of childbearing age must have a negative blood pregnancy test no later than 7 days before the first trial drug is administered.
9. Agreed to follow the experimental treatment plan and visit plan, voluntarily enrolled in the study, and signed written informed consent.

For Other Relapsed And Refractory Non-Hodgkin's Lymphoma

1. Non-hodgkin's lymphoma was confirmed by histopathology according to world Health Organization (WHO) classification of disease, and did not respond to standard treatment;
2. ECOG physical condition score 0~2;
3. Age from 18 to 70 (including boundary value), no gender limitation;
4. Life expectancy > 3 months;
5. At least one measurable lesion with a maximum diameter ≥1.5cm is present;
6. Laboratory test results must meet the following requirements (no blood components, short acting cell growth factor, albumin and other drugs are allowed to be given within 7 days before obtaining laboratory test; Long acting growth factor is not allowed in the first 14 days) :

   * Bone marrow function: Neutrophils ≥1×10E9/L, platelets ≥50×10E9/L, and hemoglobin ≥75g/L were observed without growth factor support treatment.
   * Liver function: AST and ALT ≤2×ULN (no liver invasion); Alanine aminotransferase or/and aspartate aminotransferase ≤5×ULN (liver aggressor). Total bilirubin ≤2×ULN;
   * Renal function: serum creatinine ≤2×ULN and creatinine clearance rate >50mL/min;
   * Blood coagulation function: international standardized ratio (INR) ≤1.5×ULN and activated partial thrombin time (APTT) ≤1.5×ULN;
7. Agreed to follow the experimental treatment plan and visit plan, voluntarily enrolled in the study, and signed written informed consent.

Exclusion Criteria:

* For Patients With Relapsed And Refractory CLL/SLL/PLL And Initial Treated T-PLL

  1. Central nervous system (CNS) or meningeal involvement or history of such involvement before enrollment;
  2. Received systemic steroid hormone (dose equivalent to prednisone ≥10mg/ day) and antitumor therapy within 7 days prior to initial administration of the study drug, chemotherapy, targeted therapy, radiotherapy or antibody therapy within 4 weeks or 5 half-lives, whichever is older; Failure to recover from AE associated with prior systemic antitumor therapy to nCI General Adverse Event Term version 5.0 (CT CAE Version 5.0) grade ≤1 (except hair loss);
  3. Those who had undergone major surgery, severe trauma or were expected to undergo major surgery during the study period within 4 weeks prior to the first administration of the study drug and were judged by the investigator to be unsuitable for inclusion;
  4. Autoimmune cytopenia with clinical manifestations;
  5. Have a history of active, known autoimmune deficiency, or other acquired, congenital immune deficiency diseases, or a history of organ transplantation;
  6. There was a history of other active malignant tumors within 2 years prior to the entry of the study, except for the following cases :(1) effectively controlled cervical cancer in situ; (2) effectively controlled local basal cell carcinoma of skin; (3) Other previous malignant tumors that have been clinically cured and have no clinical signs for ≥5 years;
  7. Currently has clinical significance of cardiovascular disease, activity, such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, according to the New York heart association functional class determine any 3 or 4 heart disease, or a period of 6 months before screening history of myocardial infarction, or heart left ventricular ejection fraction < 50%;
  8. Had active systemic infections (bacterial, fungal, viral, etc.) within 2 weeks prior to enrollment, including infections being treated with oral or intravenous antibiotics;
  9. Known patients with acute or chronic active hepatitis b (HBsAg positive and HBV DNA viral load ≥200IU/mL or ≥10E3 copy number /mL, other abnormal results will be determined by the investigator whether to add quantitative HBV DNA test or exclude); Acute or active hepatitis C (HCV antibody positive); And other acquired, congenital immunodeficiency diseases, including but not limited to HIV-infected persons; Or treponema pallidum antibody positive; Or CMV-DNA positive;
  10. Patients with or clinically suspected Richter's syndrome at the time of screening;
  11. Patients who received or received radiation therapy within the first 4 weeks of enrollment (except for treated bone marrow volume less than 10% and patients with evaluable lesions beyond the radiation report). Prior radioimmunotherapy within 3 months prior to initiation of the study drug;
  12. Are currently participating in an interventional clinical trial treatment, or have been treated with another clinical trial drug or device within 4 weeks prior to initial administration;
  13. Received any live virus vaccine or attenuated live vaccine within 3 months prior to enrollment;
  14. Prior allogeneic stem cell transplantation or autologous hematopoietic stem cell transplantation or any active graft-versus-host disease basis or immunosuppressant use within 21 days prior to initiation of investigational therapy;
  15. Known history of allergic diseases or severe allergies; Or is known to be allergic to protein preparations, biological agents, or any component of the test drug;
  16. Those who have a history of drug abuse or drug abuse after inquiry;
  17. Pregnant or lactating women;
  18. The investigator considered that the patient had other conditions that might affect compliance or ineligibility for the study.
* For Other Relapsed And Refractory Non-Hodgkin's Lymphoma

  1. Highly aggressive lymphoma of indolent lymphoma transformation;
  2. Known patients with acute or chronic active hepatitis b (HBsAg positive and HBV DNA viral load ≥200IU/mL or ≥10E3 copy number /mL, other abnormal results will be determined by the investigator whether to add quantitative HBV DNA test or exclude); Acute or active hepatitis C (HCV antibody positive); And other acquired, congenital immunodeficiency diseases, including but not limited to hiv-infected persons; Or treponema pallidum antibody positive; Or cmV-DNA positive;
  3. Received any anti-tumor therapy (including radiotherapy, chemotherapy, hormone therapy [dose equivalent to prednisone ≥10mg/ day], surgery or targeted therapy, immunotherapy, etc.) within 4 weeks or 5 half-life periods (whichever is longer) prior to the start of the study drug; Recovery from AE associated with prior systemic antitumor therapy to NCI General Adverse Event Term version 5.0 (CT CAE Version 5.0) grade ≤1 (except hair loss);
  4. Clinically significant heart disease, including unstable angina, acute myocardial infarction 6 months prior to randomization, congestive heart failure (NYHA) heart function grade III or IV; Or left ventricular ejection fraction < 50%;
  5. Lymphoma patients with central nervous system (CNS) invasion before enrollment;
  6. Known history of prior drug allergy; Or is known to be allergic to protein preparations, biological agents, or any component of the test drug;
  7. Those who had undergone major surgery or severe trauma within 4 weeks prior to treatment and were judged by the investigator to be unfit for inclusion;
  8. Had received autologous or allogeneic hematopoietic stem cell transplantation before enrollment;
  9. There was a history of other active malignant tumors within 2 years before entering the study, except for the following cases :(1) effectively controlled cervical cancer in situ; (2) effectively controlled local basal cell carcinoma of skin; (3) Other malignant tumors that have been clinically cured and have no clinical signs for ≥5 years;
  10. Had an active systemic infection (bacterial, fungal, viral, etc.) within 2 weeks prior to enrollment, including an infection being treated with oral or intravenous antibiotics;
  11. Participants in other clinical trials within 4 weeks prior to enrollment;
  12. Received any live virus vaccine or attenuated live vaccine within 3 months prior to enrollment;
  13. Autoimmune cytopenia with clinical manifestations;
  14. A history of drug abuse or drug abuse upon inquiry;
  15. Pregnant or lactating women;
  16. The investigator considered that the patient had other conditions that might affect compliance or ineligibility for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0 | 6 weeks
  Adverse events that occurred during the entire study period were evaluated and graded according to NCI-CTCAE v5.0, and dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) were observed.
  Safety evaluation indexes include vital signs, physical examination, 12-lead electrocardiogram, echocardiography, clinical laboratory examination indexes (blood routine, blood biochemistry, urine routine, coagulation function, etc.), changes of ECOG physical fitness score, adverse events and serious adverse event, etc.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（single administration） | 1 weeks
  Area under the plasma concentration versus time curve(AUC 0-∞)
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（single administration） | 1 weeks
  Area under the plasma concentration versus time curve(AUC 0-t）
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（single administration） | 1 weeks
  Peak Plasma Time（Tmax）
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（single administration） | 1 weeks
  Peak Plasma Concentration（Cmax）
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（single administration） | 1 weeks
  Plasma clearance（CL）
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（single administration） | 1 weeks
  Half-life of the drug（t1/2）
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  Steady State Maximum Concentration(Cmax,ss)
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  Steady State Minimal Concentration(Cmin,ss)
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  Steady State Peak Plasma Time(Tmax.ss)
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  Half-life of the drug（t1/2）
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  Steady State Area under the plasma concentration versus time curve(AUC 0-t),ss
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  fluctuation degree
Pharmacokinetic (PK) evaluation of anti-CD52 monoclone antibody（Multiple administration） | 11 weeks
  fluctuation coefficient
Efficacy evaluation of anti-CD52 monoclone antibody | 16 weeks
  ORR (including CR and PR), disease control rate (DCR), remission duration (DOR) and progression-free survival (PFS) in objective remission rate
Immunogenicity evaluation of anti-CD52 monoclone antibody | 16 weeks
  drug-resistant antibody (ADA) and neutralizing antibody (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: jianyong Li, Principal Investigator — Jiangsu Provincial People's Hospital
Locations (1):
- Jiangsu Provincial People's Hospital, Najing, Jiangsu, China